CLINICAL TRIAL: NCT04700787
Title: A Phase 1, Multi-Center, Open-Label Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Sulopenem and Sulopenem Etzadroxil + Probenecid in Adolescent Patients With Bacterial Infection
Brief Title: Safety, Tolerability, and Pharmacokinetics of Sulopenem in Adolescents
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment challenges and change in development plan necessitating a change in study design
Sponsor: Iterum Therapeutics, International Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IT001-106
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Urinary Tract Infections; Pyelonephritis Acute; Intraabdominal Infections
MeSH Terms: conditions — Urinary Tract Infections; Intraabdominal Infections | interventions — sulopenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sulopenem (Experimental): Sulopenem intravenous 1000 mg (single dose) on Day 1 followed by oral sulopenem etzadroxil/probenecid 500 mg/500 mg (single dose) on Day 2.
  Interventions: Drug: Sulopenem

INTERVENTIONS:
Drug: Sulopenem — sulopenem intravenous 1000 mg on Day 1 and then sulopenem etzadroxil/probenecid oral 500 mg/500 mg on Day 2

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of intravenous sulopenem and oral sulopenem etzadroxil/probenecid in adolescent patients.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will be screened for eligibility. Hospitalized patients who are 12-18 years of age and who are receiving background antibiotic treatment for uncomplicated urinary tract infection, complicated urinary tract infection, acute pyelonephritis, or complicated intraabdominal infection, and who meet eligibility requirements will receive a single 1000 mg IV dose of sulopenem on Day 1. The following day, patients will receive a single dose of 500 mg of sulopenem etzadroxil and 500 mg of probenecid given orally as a bilayer tablet. During treatment, pharmacokinetic samples will be collected and patients will be monitored for safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's parent/both parents or guardian must provide written informed consent and a statement of assent from the adolescent patient (if required by Institutional Review Board [IRB] according to local regulations and guidelines) must be obtained prior to any study-related procedures.
2. Patient is male or female adolescent who are ≥12 and <18 years of age.
3. Patient has a diagnosis of uUTI, cUTI, AP, or cIAI as documented by the treating physician
4. Patient will be hospitalized for urinary tract infection, acute pyelonephritis, or complicated intraabdominal infection for at least 48 hours and be receiving appropriate anti-infective treatment.
5. Patient must have sufficient venous access to permit administration of study drug, collection of PK samples, and monitoring of laboratory safety variables.
6. Female patients who are post-menarche must not be pregnant or breast feeding and must have a documented negative serum pregnancy test at Screening.
7. Post-menarchal females and post-pubertal males must agree to use a highly effective method of birth control with partners of childbearing potential throughout the duration of the study and for 1 month following the last dose of study drug.
8. Patient must be willing to follow all study procedures.

Exclusion Criteria:

1. Patient has creatinine clearance <90 mL/min using the Cockcroft-Gault formula.
2. Patient is unable to tolerate oral medications.
3. Patient has presence of Endocarditis, Meningitis, Necrotizing fasciitis, or Gas gangrene
4. Patient has signs of severe sepsis
5. Patient has evidence of active liver disease or hepatic dysfunction
6. Patient has neutropenia with absolute neutrophil count <500 cells/mm3.
7. Patient has history of solid organ transplantation reported at any time.
8. Patient has any finding that, in the view of the Investigator, would compromise the patient's safety requirements.
9. Patient has known allergies to penicillin, carbapenems, and/or cephalosporins, known allergy to probenecid, or severe allergic reactions to any drug in the past.
10. Patient has history of intolerance to β-lactam antibiotics, including but not limited to a history of clinically significant diarrhea/loose stools.
11. Patient has a history of hypersensitivity to the study drug or any of the excipients or to medicinal products with similar chemical structures.
12. Patient has involvement in the planning and/or conduct of this study
13. Patient has participated in any other clinical study where an investigational product was ingested within 30 days or 5 half-lives of the drug (whichever is longer) prior to the current study.
14. Patient has definite or suspected personal history or family history of clinically significant adverse drug reactions.
15. Patient has history or presence of GI, hepatic, or renal disease, or other conditions known to interfere with absorption, distribution, metabolism, or excretion of drugs.
16. Patient had treatment in the previous 3 months with any drug known to have a well-defined potential for hepatotoxicity (eg, halothane).
17. Patient weighs <35 kg.
18. Patient is pregnant or lactating.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration | To be measured at 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 8.0, 9.0, 10.0, and 12.0 hours post dose
  Maximum plasma concentration (Cmax) of sulopenem at multiple timepoints after dose

SECONDARY OUTCOMES:
Time to maximum plasma concentration | To be measured at 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 8.0, 9.0, 10.0, and 12.0 hours post dose
  Time to maximum plasma concentration (Tmax) of sulopenem at multiple timepoints after dose
Time above minimum inhibitory concentration | To be measured at 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 8.0, 9.0, 10.0, and 12.0 hours post dose
  Time above minimum inhibitory concentration (MIC) at multiple timepoints after dose
Area under the plasma concentration-time curve from time zero to time of last quantifiable plasma concentration | To be measured at 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 8.0, 9.0, 10.0, and 12.0 hours post dose
  Area under the plasma concentration-time curve (AUC) from time zero to time of last quantifiable plasma concentration at multiple timepoints after dose
Area under the plasma concentration-time curve from time zero extrapolated to infinity | To be measured at 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 8.0, 9.0, 10.0, and 12.0 hours post dose
  Area under the plasma concentration-time curve (AUC) from time zero extrapolated to infinity at multiple timepoints after dose
Percentage of area under the concentration-time curve extrapolated | To be measured at 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 8.0, 9.0, 10.0, and 12.0 hours post dose
  Percentage of area under the concentration-time curve (AUC) extrapolated at multiple timepoints after dose
Terminal elimination half-life | To be measured at 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 8.0, 9.0, 10.0, and 12.0 hours post dose
  Terminal elimination half-life at multiple timepoints after dose
Total body clearance for intravenous administration | To be measured at 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 8.0, 9.0, 10.0, and 12.0 hours post dose
  Total body clearance for intravenous administration at multiple timepoints after intravenous dose
Apparent total body clearance for oral administration | To be measured at 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 8.0, 9.0, 10.0, and 12.0 hours post dose
  Apparent total body clearance for oral administration at multiple timepoints after oral dose
Volume of distribution for intravenous administration | To be measured at 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 8.0, 9.0, 10.0, and 12.0 hours post dose
  Volume of distribution for intravenous administration at multiple timepoints after intravenous dose
Apparent volume of distribution for oral administration | To be measured at 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 8.0, 9.0, 10.0, and 12.0 hours post dose
  Apparent volume of distribution for oral administration at multiple timepoints after oral dose

CONTACTS AND LOCATIONS:
Overall Officials: Steven I Aronin, MD, Study Director — Employee
Locations (1):
- Medical Facility, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No